CLINICAL TRIAL: NCT05937828
Title: "French National Cohort of Patients With Pediatric-onset of Autoimmune Cytopenia (OBS'CEREVANCE Cohort)"
Brief Title: OBS'CEREVANCE: French Cohort of Pediatric Autoimmune Cytopenia
Acronym: OBS'CEREVANCE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/08
Record Dates: First submitted 2023-03-14; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Immune Thrombocytopenia; Autoimmune Hemolytic Anemia; Evans Syndrome
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Anemia, Hemolytic, Autoimmune; Evans Syndrome | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 19 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Immune thrombocytopenia (ITP): Immune thrombocytopenia (ITP) : defined according to the international working group criteria (Rodeghiero et al., Blood 2009).
  Interventions: Other: data collection
- Autoimmune Hemolytic anemia (AIHA): Autoimmune haemolytic anaemia (AIHA) : Hb < 110 g/L with a positive direct antiglobulin test (DAT) and at least one of the following haemolysis criteria: reticulocyte count > 120 G/L, free bilirubin > 17 mmol/L, or haptoglobin < 10 mg/dL.
  Interventions: Other: data collection
- Evans syndrome (all bi or tri cytopenias): Evans syndrome (ES) : simultaneous (less than 1 month) or sequential association of at least two autoimmune cytopenia among ITP, AIHA and autoimmune neutropenia (AIN).
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — description of the long-term health of adult patients, identification of the heterogenous genetic underlying pathophysiologic contexts, study of the benefit-risk balance of treatments, including the growing development of targeted therapies.

SUMMARY:
From 2004, OBS'CEREVANCE is a national real-world prospective clinical cohort of patients with auto-immune cytopenia of pediatric-onset : Immune thrombocytopenia (ITP), Autoimmune Hemolytic anemia (AIHA), or Evans syndrome (all bi or tri cytopenias). Thanks to the collaboration of the 30 French pediatric hematologic centers, this cohort supports all of the Rare Disease Centre CEREVANCE (Centre de Référence National des Cytopénies Auto-Immunes de l'Enfant) missions for care, education and research. Specifically, this original unbiased database allows to describe the long-term health of adult patients, to identify the heterogenous genetic underlying pathophysiologic contexts, and to study the benefit-risk balance of treatments, including the growing development of targeted therapies.

DETAILED DESCRIPTION:
Immune thrombocytopenic purpura (ITP) and autoimmune hemolytic anemia (AHAI) are rare childhood diseases that involve autoimmune destruction of platelets and erythrocytes respectively.

They may be associated with an even rarer entity, Evans syndrome (ES). These three conditions are referred to as autoimmune cytopenias (AIC).

In association with CAI, patients may present with various immunopathological (IM) manifestations such as lymphoproliferation, autoimmune autoimmune/autoinflammatory organ diseases that may be absent at the time of at the time of diagnosis of CAI and develop during follow-up.

Since 2004, the CEREVANCE reference center for childhood autoimmune CEREVANCE has been coordinating a national prospective cohort of patients with pediatric-onset CAI including over 1900 patients (data 05/2023).

Thanks to the collaboration of the 30 French pediatric hematologic centers, this cohort supports all of the Rare Disease Centre CEREVANCE (Centre de Référence National des Cytopénies Auto-Immunes de l'Enfant) missions for care, education and research. Specifically, this original unbiased database allows to describe the long-term health of adult patients, to identify the heterogenous genetic underlying pathophysiologic contexts, and to study the benefit-risk balance of treatments, including the growing development of targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ITP, AIHA, Evans Syndrome
* Onset before the age of 18

Exclusion Criteria:

* Opposition of legal representative or to data collection

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Each of the 30 hemato-immunologic pediatric unit in France guaranties the prospective in real time inclusion in the cohort of all the children diagnosed in their unit, before 18 years old, with ITP, AIHA or Evans syndrome diagnosis, whatever the date of diagnosis at the date of inclusion.
  This observational cohort is prospective from the day of initial diagnosis of the auto-immune cytopenia The pediatricians from this rare disease CEREVANCE national network follow national guidelines for evaluation and treatment (PNDS 2009, 2017)
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2010-09-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
AIC context | Baseline
  Number of patients with immunopathological manifestations (IM), systemic erythematosus lupus (SLE), primary immunodeficiency (PID).

SECONDARY OUTCOMES:
Treatment lines | every 6 months after baseline up to 19 years
  Percentage of patients with each treatment by line of treatments
Adverse drug reactions | every 6 months after baseline up to 19 years
  Percentage of patients with adverse drug reaction reported by investigators
Events | every 6 months after baseline up to 19 years
  Percentage of patients with other events of interest like cancer, infection, thrombosis, death
AIC context | every 6 months after baseline up to 19 years
  Number of patients with immunopathological manifestations (IM), systemic erythematosus lupus (SLE), primary immunodeficiency (PID).

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie ALADJIDI, MD, Principal Investigator — University Hospital, Bordeaux
Locations (9):
- France (9):
  - CHU Amiens Picardie Service d' Onco-Immuno-Hématologie Pédiatrique, Amiens
  - CHU d'Angers Unité d'Hémato-Oncologie Pédiatrique, Angers
  - BESANCON CHU de Besançon Hôpital Jean MINJOZ Unité d'Hémato-Oncologie Pédiatrique, Pédiatrie 1, Besançon
  - CHU de Bordeaux - Unité d'Hématologie et d'Oncologie pédiatrique, Bordeaux
  - CHU BREST Hôpital Morvan Unité d'Onco-Hématologie, Brest
  - CHU de Caen Unité d'Onco-Hématologie, Caen
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - APHP Hôpital Bicêtre Service de Pédiatrie générale, Paris
  - CH de Cornouaille Service de Pédiatrie, Quimper

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ducassou S, Leverger G, Fernandes H, Chambost H, Bertrand Y, Armari-Alla C, Nelken B, Monpoux F, Guitton C, Leblanc T, Fisher A, Lejars O, Jeziorski E, Fouissac F, Lutz P, Pasquet M, Pellier I, Piguet C, Vic P, Bayart S, Marie-Cardine A, Michel M, Perel Y, Aladjidi N. Benefits of rituximab as a second-line treatment for autoimmune haemolytic anaemia in children: a prospective French cohort study. Br J Haematol. 2017 Jun;177(5):751-758. doi: 10.1111/bjh.14627. Epub 2017 Apr 26. PMID 28444729
- [Background] Aladjidi N, Jutand MA, Beaubois C, Fernandes H, Jeanpetit J, Coureau G, Gilleron V, Kostrzewa A, Lauroua P, Jeanne M, Thiebaut R, Leblanc T, Leverger G, Perel Y. Reliable assessment of the incidence of childhood autoimmune hemolytic anemia. Pediatr Blood Cancer. 2017 Dec;64(12). doi: 10.1002/pbc.26683. Epub 2017 Jul 27. PMID 28748541
- [Background] Penel Page M, Bertrand Y, Fernandes H, Kherfellah D, Leverger G, Leblanc T, Libbrecht C, Michel G, Jeziorski E, Armari-Alla C, Nelken B, Pellier I, Pasquet M, Perel Y, Aladjidi N. Treatment with cyclosporin in auto-immune cytopenias in children: The experience from the French cohort OBS'CEREVANCE. Am J Hematol. 2018 May 14. doi: 10.1002/ajh.25137. Online ahead of print. No abstract available. PMID 29756344
- [Background] Pincez T, Neven B, Le Pointe HD, Varlet P, Fernandes H, Gareton A, Leverger G, Leblanc T, Chambost H, Michel G, Pasquet M, Millot F, Hermine O, Mathian A, Hully M, Zephir H, Hamidou M, Durand JM, Perel Y, Landman-Parker J, Rieux-Laucat F, Aladjidi N. Neurological Involvement in Childhood Evans Syndrome. J Clin Immunol. 2019 Feb;39(2):171-181. doi: 10.1007/s10875-019-0594-3. Epub 2019 Jan 22. PMID 30671780
- [Background] Hadjadj J, Aladjidi N, Fernandes H, Leverger G, Magerus-Chatinet A, Mazerolles F, Stolzenberg MC, Jacques S, Picard C, Rosain J, Fourrage C, Hanein S, Zarhrate M, Pasquet M, Abou Chahla W, Barlogis V, Bertrand Y, Pellier I, Colomb Bottollier E, Fouyssac F, Blouin P, Thomas C, Cheikh N, Dore E, Pondarre C, Plantaz D, Jeziorski E, Millot F, Garcelon N, Ducassou S, Perel Y, Leblanc T, Neven B, Fischer A, Rieux-Laucat F; members of the French Reference Center for Pediatric Autoimmune Cytopenia (CEREVANCE). Pediatric Evans syndrome is associated with a high frequency of potentially damaging variants in immune genes. Blood. 2019 Jul 4;134(1):9-21. doi: 10.1182/blood-2018-11-887141. Epub 2019 Apr 2. PMID 30940614
- [Background] Margot H, Boursier G, Duflos C, Sanchez E, Amiel J, Andrau JC, Arpin S, Brischoux-Boucher E, Boute O, Burglen L, Caille C, Capri Y, Collignon P, Conrad S, Cormier-Daire V, Delplancq G, Dieterich K, Dollfus H, Fradin M, Faivre L, Fernandes H, Francannet C, Gatinois V, Gerard M, Goldenberg A, Ghoumid J, Grotto S, Guerrot AM, Guichet A, Isidor B, Jacquemont ML, Julia S, Khau Van Kien P, Legendre M, Le Quan Sang KH, Leheup B, Lyonnet S, Magry V, Manouvrier S, Martin D, Morel G, Munnich A, Naudion S, Odent S, Perrin L, Petit F, Philip N, Rio M, Robbe J, Rossi M, Sarrazin E, Toutain A, Van Gils J, Vera G, Verloes A, Weber S, Whalen S, Sanlaville D, Lacombe D, Aladjidi N, Genevieve D. Immunopathological manifestations in Kabuki syndrome: a registry study of 177 individuals. Genet Med. 2020 Jan;22(1):181-188. doi: 10.1038/s41436-019-0623-x. Epub 2019 Jul 31. PMID 31363182
- [Background] Ducassou S, Gourdonneau A, Fernandes H, Leverger G, Pasquet M, Fouyssac F, Bayart S, Bertrand Y, Michel G, Jeziorski E, Thomas C, Abouchallah W, Viard F, Guitton C, Cheikh N, Pellier I, Carausu L, Droz C, Leblanc T, Aladjidi N; Centre de Reference National des Cytopenies Auto-immunes de l'Enfant (CEREVANCE). Second-line treatment trends and long-term outcomes of 392 children with chronic immune thrombocytopenic purpura: the French experience over the past 25 years. Br J Haematol. 2020 Jun;189(5):931-942. doi: 10.1111/bjh.16448. Epub 2020 Mar 4. PMID 32130726
- [Background] Ducassou S, Fernandes H, Savel H, Bertrand Y, Leblanc T, Abou Chahla W, Pasquet M, Leverger G, Barlogis V, Thomas C, Bayart S, Pellier I, Armari-Alla C, Guitton C, Cheikh N, Kherfellah D, Vassal G, Thiebaut R, Laghouati S, Aladjidi N. Prospective Evaluation of the First Option, Second-Line Therapy in Childhood Chronic Immune Thrombocytopenia: Splenectomy or Immunomodulation. J Pediatr. 2021 Apr;231:223-230. doi: 10.1016/j.jpeds.2020.12.018. Epub 2020 Dec 17. PMID 33340549
- [Background] Pincez T, Fernandes H, Leblanc T, Michel G, Barlogis V, Bertrand Y, Neven B, Chahla WA, Pasquet M, Guitton C, Marie-Cardine A, Pellier I, Armari-Alla C, Benadiba J, Blouin P, Jeziorski E, Millot F, Paillard C, Thomas C, Cheikh N, Bayart S, Fouyssac F, Piguet C, Deparis M, Briandet C, Dore E, Picard C, Rieux-Laucat F, Landman-Parker J, Leverger G, Aladjidi N. Long term follow-up of pediatric-onset Evans syndrome: broad immunopathological manifestations and high treatment burden. Haematologica. 2022 Feb 1;107(2):457-466. doi: 10.3324/haematol.2020.271106. PMID 33440924
- [Background] Pincez T, Aladjidi N, Heritier S, Garnier N, Fahd M, Abou Chahla W, Fernandes H, Dichamp C, Ducassou S, Pasquet M, Bayart S, Moshous D, Cheikh N, Paillard C, Plantaz D, Jeziorski E, Thomas C, Guitton C, Deparis M, Marie Cardine A, Stephan JL, Pellier I, Dore E, Benadiba J, Pluchart C, Briandet C, Barlogis V, Leverger G, Leblanc T. Determinants of long-term outcomes of splenectomy in pediatric autoimmune cytopenias. Blood. 2022 Jul 21;140(3):253-261. doi: 10.1182/blood.2022015508. PMID 35443028
- [Background] Pincez T, Fernandes H, Pasquet M, Abou Chahla W, Granel J, Heritier S, Fahd M, Ducassou S, Thomas C, Garnier N, Barlogis V, Jeziorski E, Bayart S, Chastagner P, Cheikh N, Guitton C, Paillard C, Lejeune J, Millot F, Li-Thiao Te V, Mallebranche C, Pellier I, Neven B, Armari-Alla C, Carausu L, Piguet C, Benadiba J, Pluchart C, Stephan JL, Deparis M, Briandet C, Dore E, Marie-Cardine A, Leblanc T, Leverger G, Aladjidi N. Impact of age at diagnosis, sex, and immunopathological manifestations in 886 patients with pediatric chronic immune thrombocytopenia. Am J Hematol. 2023 Jun;98(6):857-868. doi: 10.1002/ajh.26900. Epub 2023 Mar 21. PMID 36882195
- [Derived] Granel J, Fernandes H, Bader-Meunier B, Guth A, Richer O, Pillet P, Leverger G, Ducassou S, Fahd M, Pasquet M, Garnier N, Barlogis V, Guitton C, Jeziorski E, Thomas C, Bayart S, Cheikh N, Paillard C, Abou Chahla W, Chastagner P, Neven B, Millot F, Lejeune J, Li-Thiao Te V, Armari-Alla C, Briandet C, Carausu L, Deparis M, Piguet C, Benadiba J, Marie-Cardine A, Stephan JL, Pellier I, Pluchart C, Dore E, Michaux K, Heritier S, Leblanc T, Aladjidi N. Antinuclear antibody-associated autoimmune cytopenia in childhood is a risk factor for systemic lupus erythematosus. Blood. 2024 Apr 18;143(16):1576-1585. doi: 10.1182/blood.2023021884. PMID 38227934